CLINICAL TRIAL: NCT01891188
Title: Using Near-infrared Spectroscopy (NIRS) Monitor to Noninvasively Evaluate Hepatic Venous Saturation
Status: Completed | Type: Observational
Sponsor: Phoenix Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PHNX-hNIRS-12-120
Record Dates: First submitted 2012-11-30; First posted 2013-07-03 (Estimated); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Congenital Heart Disease; Arrhythmia
Keywords: hepatic blood,; cardiac cath,; hepatic oxygenation,; pediatrics
MeSH Terms: conditions — Heart Defects, Congenital; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cardiac Cath: All pediatric patients requiring cardiac catheterization who consent

SUMMARY:
Clinical studies are required to validate the hepatic NIRS monitor with other regional and global hemodynamic parameters and to evaluate its clinical use for continuous non-invasive hemodynamic monitoring. Using newer NIRS sensors the correlation between hepatic regional oxygen saturation and hepatic venous oxygen saturation (SvHO2) needs to be determined. If found to correlate then the NIRS can be used to evaluate early liver transplant failure and/or hepatic artery thrombosis, used as an early marker for shock, and necrotizing enterocolitis, and finally used in the outpatient setting to evaluate patients with chronic liver pathologies. If our validation study finds that NIRS monitors are an appropriate marker of hepatic venous saturation then it will lead to further clinical studies.

ELIGIBILITY:
Inclusion Criteria:

* All pediatric patients (0-18yrs) undergoing cardiac catheterization by the participating interventional cardiologist at Phoenix Children's Hospital will be recruited for this investigation

Exclusion Criteria:

* emergency catheterizations,
* procedures in hemodynamically unstable patients,
* patients with repeat catheterizations that have already enrolled in the study

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All pediatric patients (0-18yrs) undergoing cardiac catheterization by the participating interventional cardiologist at Phoenix Children's Hospital will be recruited for this investigation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2016-07-01 (Actual)

PRIMARY OUTCOMES:
Degree of Hepatic Venous Saturation using NIRS | 5 minutes
  The investigators strive to discover a noninvasive measure of hepatic venous saturation. The use of NIRS monitoring for global oxygen saturation has been used in the inpatient population. This project aims to use hepatic NIRS monitor as a surrogate marker for hepatic and splanchnic oxygenation.

CONTACTS AND LOCATIONS:
Overall Officials: Rohit Rao, MD, Principal Investigator — Phoenix Children's Hospital
Locations (1):
- Phoenix Children's Hospital, Phoenix, Arizona, United States

REFERENCES:
- [Background] FDA 510K Clearances. (2001) Somanetics Corp Adult/Pediatric Cerebral Oximeter Model 5100.http://www.fda.gov/MedicalDevices/ProductsandMedicalProcedures/DeviceApprovalsandClearances/510kClearances/ucm093461.htm
- [Background] Marin T, Moore J. Understanding near-infrared spectroscopy. Adv Neonatal Care. 2011 Dec;11(6):382-8. doi: 10.1097/ANC.0b013e3182337ebb. PMID 22123468
- [Background] Hayashida M, Kin N, Tomioka T, Orii R, Sekiyama H, Usui H, Chinzei M, Hanaoka K. Cerebral ischaemia during cardiac surgery in children detected by combined monitoring of BIS and near-infrared spectroscopy. Br J Anaesth. 2004 May;92(5):662-9. doi: 10.1093/bja/aeh120. Epub 2004 Mar 19. PMID 15033888
- [Background] Hoffman GM, Stuth EA, Jaquiss RD, Vanderwal PL, Staudt SR, Troshynski TJ, Ghanayem NS, Tweddell JS. Changes in cerebral and somatic oxygenation during stage 1 palliation of hypoplastic left heart syndrome using continuous regional cerebral perfusion. J Thorac Cardiovasc Surg. 2004 Jan;127(1):223-33. doi: 10.1016/j.jtcvs.2003.08.021. PMID 14752434
- [Background] Nollert G, Jonas RA, Reichart B. Optimizing cerebral oxygenation during cardiac surgery: a review of experimental and clinical investigations with near infrared spectrophotometry. Thorac Cardiovasc Surg. 2000 Aug;48(4):247-53. doi: 10.1055/s-2000-6895. PMID 11005605
- [Background] Watzman HM, Kurth CD, Montenegro LM, Rome J, Steven JM, Nicolson SC. Arterial and venous contributions to near-infrared cerebral oximetry. Anesthesiology. 2000 Oct;93(4):947-53. doi: 10.1097/00000542-200010000-00012. PMID 11020744
- [Background] Wyatt JS, Cope M, Delpy DT, Wray S, Reynolds EO. Quantification of cerebral oxygenation and haemodynamics in sick newborn infants by near infrared spectrophotometry. Lancet. 1986 Nov 8;2(8515):1063-6. doi: 10.1016/s0140-6736(86)90467-8. PMID 2877225
- [Background] Yoshitani K, Kawaguchi M, Iwata M, Sasaoka N, Inoue S, Kurumatani N, Furuya H. Comparison of changes in jugular venous bulb oxygen saturation and cerebral oxygen saturation during variations of haemoglobin concentration under propofol and sevoflurane anaesthesia. Br J Anaesth. 2005 Mar;94(3):341-6. doi: 10.1093/bja/aei046. Epub 2004 Dec 10. PMID 15591331
- [Background] Petros AJ, Heys R, Tasker RC, Fortune PM, Roberts I, Kiely E. Near infrared spectroscopy can detect changes in splanchnic oxygen delivery in neonates during apnoeic episodes. Eur J Pediatr. 1999 Feb;158(2):173-4. doi: 10.1007/s004310051046. No abstract available. PMID 10048622
- [Background] Nagdyman N, Fleck T, Barth S, Abdul-Khaliq H, Stiller B, Ewert P, Huebler M, Kuppe H, Lange PE. Relation of cerebral tissue oxygenation index to central venous oxygen saturation in children. Intensive Care Med. 2004 Mar;30(3):468-71. doi: 10.1007/s00134-003-2101-8. Epub 2004 Jan 13. PMID 14722637
- [Background] Schulz G, Weiss M, Bauersfeld U, Teller J, Haensse D, Bucher HU, Baenziger O. Liver tissue oxygenation as measured by near-infrared spectroscopy in the critically ill child in correlation with central venous oxygen saturation. Intensive Care Med. 2002 Feb;28(2):184-9. doi: 10.1007/s00134-001-1182-5. Epub 2002 Jan 12. PMID 11907662
- [Background] Weiss M, Dullenkopf A, Kolarova A, Schulz G, Frey B, Baenziger O. Near-infrared spectroscopic cerebral oxygenation reading in neonates and infants is associated with central venous oxygen saturation. Paediatr Anaesth. 2005 Feb;15(2):102-9. doi: 10.1111/j.1460-9592.2005.01404.x. PMID 15675925
- [Background] Nollert G, Mohnle P, Tassani-Prell P, Uttner I, Borasio GD, Schmoeckel M, Reichart B. Postoperative neuropsychological dysfunction and cerebral oxygenation during cardiac surgery. Thorac Cardiovasc Surg. 1995 Oct;43(5):260-4. doi: 10.1055/s-2007-1013224. PMID 8610284
- [Background] Berens RJ, Stuth EA, Robertson FA, Jaquiss RD, Hoffman GM, Troshynski TJ, Staudt SR, Cava JR, Tweddell JS, Bert Litwin S. Near infrared spectroscopy monitoring during pediatric aortic coarctation repair. Paediatr Anaesth. 2006 Jul;16(7):777-81. doi: 10.1111/j.1460-9592.2006.01956.x. PMID 16879521
- [Background] Tsuji M, Saul JP, du Plessis A, Eichenwald E, Sobh J, Crocker R, Volpe JJ. Cerebral intravascular oxygenation correlates with mean arterial pressure in critically ill premature infants. Pediatrics. 2000 Oct;106(4):625-32. doi: 10.1542/peds.106.4.625. PMID 11015501
- [Background] Beilman GJ, Groehler KE, Lazaron V, Ortner JP. Near-infrared spectroscopy measurement of regional tissue oxyhemoglobin saturation during hemorrhagic shock. Shock. 1999 Sep;12(3):196-200. doi: 10.1097/00024382-199909000-00005. PMID 10485597
- [Background] Rhee P, Langdale L, Mock C, Gentilello LM. Near-infrared spectroscopy: continuous measurement of cytochrome oxidation during hemorrhagic shock. Crit Care Med. 1997 Jan;25(1):166-70. doi: 10.1097/00003246-199701000-00030. PMID 8989194
- [Background] Yang W, Hafez T, Thompson CS, Mikhailidis DP, Davidson BR, Winslet MC, Seifalian AM. Direct measurement of hepatic tissue hypoxia by using a novel tcpO2/pCO2 monitoring system in comparison with near-infrared spectroscopy. Liver Int. 2003 Jun;23(3):163-70. doi: 10.1034/j.1600-0676.2003.00818.x. PMID 12955879
- [Background] El-Desoky AE, Jiao LR, Havlik R, Habib N, Davidson BR, Seifalian AM. Measurement of hepatic tissue hypoxia using near infrared spectroscopy: comparison with hepatic vein oxygen partial pressure. Eur Surg Res. 2000;32(4):207-14. doi: 10.1159/000008766. PMID 11014921
- [Background] El-Desoky AE, Seifalian AM, Davidson BR. Effect of graded hypoxia on hepatic tissue oxygenation measured by near infrared spectroscopy. J Hepatol. 1999 Jul;31(1):71-6. doi: 10.1016/s0168-8278(99)80165-2. PMID 10424285
- [Background] Teller J, Wolf M, Keel M, Bucher HU, Fanconi S, Baenziger O. Can near infrared spectroscopy of the liver monitor tissue oxygenation? Eur J Pediatr. 2000 Jul;159(7):549. doi: 10.1007/s004310051334. PMID 10923236
- [Background] Weiss M, Schulz G, Teller I, Dullenkopf A, Kolarova A, Sailer H, Dillier CM, Bucher HU, Gerber AC, Baenziger O. Tissue oxygenation monitoring during major pediatric surgery using transcutaneous liver near infrared spectroscopy. Paediatr Anaesth. 2004 Dec;14(12):989-95. doi: 10.1111/j.1460-9592.2004.01362.x. PMID 15601347
- [Background] Weiss M, Schulz G, Fasnacht M, Balmer C, Fischer JE, Gerber AC, Bucher HU, Baenziger O. Transcutaneously measured near-infrared spectroscopic liver tissue oxygenation does not correlate with hepatic venous oxygenation in children. Can J Anaesth. 2002 Oct;49(8):824-9. doi: 10.1007/BF03017416. PMID 12374712
- [Background] Teller J, Schwendener K, Wolf M, Keel M, Bucher HU, Fanconi S, Baenziger O. Continuous monitoring of liver oxygenation with near infrared spectroscopy during naso-gastric tube feeding in neonates. Schweiz Med Wochenschr. 2000 May 6;130(18):652-6. PMID 10846757
- [Background] Ceppa EP, Fuh KC, Bulkley GB. Mesenteric hemodynamic response to circulatory shock. Curr Opin Crit Care. 2003 Apr;9(2):127-32. doi: 10.1097/00075198-200304000-00008. PMID 12657975
- [Background] Kinoshita G, Washizu M, Motoyoshi S, Breznock EM. Effects of hypovolemic shock and reperfusion on liver blood flow in the dog. J Vet Med Sci. 1995 Aug;57(4):703-8. doi: 10.1292/jvms.57.703. PMID 8519902
- [Background] Lautt WW. The 1995 Ciba-Geigy Award Lecture. Intrinsic regulation of hepatic blood flow. Can J Physiol Pharmacol. 1996 Mar;74(3):223-33. PMID 8773400
- [Background] Lautt WW, McQuaker JE. Maintenance of hepatic arterial blood flow during hemorrhage is mediated by adenosine. Can J Physiol Pharmacol. 1989 Sep;67(9):1023-8. doi: 10.1139/y89-161. PMID 2598127
- [Background] Jakob SM, Tenhunen JJ, Laitinen S, Heino A, Alhava E, Takala J. Effects of systemic arterial hypoperfusion on splanchnic hemodynamics and hepatic arterial buffer response in pigs. Am J Physiol Gastrointest Liver Physiol. 2001 May;280(5):G819-27. doi: 10.1152/ajpgi.2001.280.5.G819. PMID 11292589
- [Background] Eipel C, Abshagen K, Vollmar B. Regulation of hepatic blood flow: the hepatic arterial buffer response revisited. World J Gastroenterol. 2010 Dec 28;16(48):6046-57. doi: 10.3748/wjg.v16.i48.6046. PMID 21182219
- [Background] Ortmann LA, Fontenot EE, Seib PM, Eble BK, Brown R, Bhutta AT. Use of near-infrared spectroscopy for estimation of renal oxygenation in children with heart disease. Pediatr Cardiol. 2011 Aug;32(6):748-53. doi: 10.1007/s00246-011-9960-5. Epub 2011 Mar 29. PMID 21445607